CLINICAL TRIAL: NCT00779168
Title: A Phase Ib Trial of Mushroom Powder in Biochemically Recurrent Prostate Cancer
Brief Title: White Button Mushroom Extract in Treating Patients With Recurrent Prostate Cancer After Local Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08012; P30CA033572 (NIH); CHNMC-08012; CDR0000617012 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flow Cytometry; Immunologic Techniques; Gas Chromatography-Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive white button mushroom extract PO twice daily on days 1-28. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: white button mushroom extract; Other: flow cytometry; Other: immunologic technique; Other: laboratory biomarker analysis; Other: gas chromatography-mass spectrometry; Other: pharmacological study

INTERVENTIONS:
Drug: white button mushroom extract — For this dose escalation study 6 patients will be treated at each of the following dosages: 4 grams PO daily, 6 grams PO daily, 8 grams PO daily, 10 grams PO daily, 12 grams PO daily and 14 grams PO daily.
Other: flow cytometry — Immune cell subset number will be evaluated by flow cytometry on blood samples collected on days -14, -7, 1, 15, 29, 57, 85 from treatment and when coming off study.
Other: immunologic technique — Testing will be performed on blood samples collected on days -14, -7, 1, 15, 29, 57, 85 from treatment and when coming off study.
Other: laboratory biomarker analysis — Performed on blood samples collected pre-study (within 4 weeks of registration) and during weeks 3, 5, 9, 13, every 4 weeks beyond week 13 and at off study.
Other: gas chromatography-mass spectrometry — Gas Chromatography-Mass Spectrometry (GC-MS) will be used to evaluate C-18 unsaturated fatty acids (CUFA) in blood samples collected on days -14, -7 prior to start of treatment. On day 1 of week 1 blood will be drawn at pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, and 6 hours post-dose and subsequently on days 15, 29, 57 and 85 and when coming off study.
Other: pharmacological study — Evaluation of C-18 unsaturated fatty acids (CUFA) in blood samples collected on days -14, -7 prior to start of treatment. On day 1 of week 1 blood will be drawn at pre-dose, 0.25, 0.5, 0.75, 1, 2, 4, and 6 hours post-dose and subsequently on days 15, 29, 57 and 85 and when coming off study.

SUMMARY:
RATIONALE: White button mushroom extract may stop or delay the development of recurrent prostate cancer.

PURPOSE: This phase I trial is studying the side effects and best dose of white button mushroom extract in treating patients with recurrent prostate cancer after local therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility and toxicity of prolonged white button mushroom extract therapy at six different dose levels in patients with biochemically recurrent prostate cancer after local therapy.

Secondary

* To analyze the effect of this regimen on a variety of biomarkers including testosterone, dihydrotestosterone, dehydroepiandrosterone, estrogens, aromatase, parameters of immune function, and circulating tumor cells.
* To assess the effect of this regimen on PSA kinetics as a measure of disease activity in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral white button mushroom extract twice daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Blood and urine samples are collected periodically for pharmacokinetic, pharmacodynamic, and immunologic correlative studies. Plasma and urine samples are analyzed for quantification of conjugated unsaturated fatty acids via gas chromatography-mass spectometry. Plasma samples are analyzed for inhibition of aromatase via aromatase activity analysis and the effect of treatment on immune cytokines levels via immunobiologic assays. Peripheral blood mononuclear cells are analyzed for the effect of treatment on immune cell subsets and NK cell function via multi-parameter flow cytometry; effect of treatment on NK cell activation status via staining method; and measurement of circulating tumor cells via fluorescence microscopy, fiber-optic array scanning technology (FAST), or high-speed flow cytometry. Additional serum samples are collected for future studies.

Patients complete a diary listing days of administration of treatment and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically or cytologically confirmed history of adenocarcinoma of the prostate Patients must have a PSA failure defined as PSA of >= 0.2 ng/ml that has increased above nadir following prostatectomy If radiation or other local therapy was used as a primary therapy and no prostatectomy was performed patients must have PSA increase of 2.0 above post-therapy nadir; PSA value must be increasing based on two consecutive measurements each separated by at least 2 weeks with no clinical or radiographic evidence of metastatic disease; PSA values that meet the criteria for eligibility within 4 weeks of registration are acceptable to document eligibility for enrollment on this study; PSA level obtained after registration and prior to the first course will be used as the "baseline" PSA as per the schema but will not determine eligibility for participation
* Patients must have had at least three PSA measurements over a minimum of three months available prior to enrollment to this study
* Patients may have received any number of local therapies (radical prostatectomy, external beam radiation therapy, radioactive seed implantation, cryotherapy)
* Bone scan and computed tomography (CT) scan of the chest, abdomen and pelvis negative for metastatic disease within 2 months prior to registration
* Patients must have a performance status of 0, 1, or 2
* All patients will have malignancy confirmed by review of their biopsy specimens by the Division of Pathology, City of Hope National Medical Center; if no pathological specimen is available for review, the patient may still be included if the patient has clearly documented prostate cancer per pathology report and a specimen request is documented as having been made for tissue from the outside facility but a specimen was unable to be obtained
* Serum creatinine =< 2.5 mg/dL
* Baseline liver function tests including bilirubin =< 1.5 x the institutional upper limit of normal and serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) =< 2.5 x the institutional upper limit of normal
* White blood cells (WBC) >= 2000
* Platelets >= 50,000

Exclusion Criteria:

* Patients with evidence of metastatic disease
* PSA progression not verified by sequential rising PSA as discussed in the eligibility section
* Patients who have received prior cytotoxic chemotherapy or androgen ablative therapy for recurrent disease
* Patients currently receiving biological response modifiers, or corticosteroids
* Patients are permitted to have received up to 24 months of neoadjuvant or adjuvant hormone ablation in conjunction with their primary definitive therapy; androgen deprivation must have been completed at least 6 months prior to registration and testosterone level must be > 50; no complementary or alternative therapy (e.g. St. John's Wort, PC-SPES, or other herbal remedies taken for the purpose of treating prostate cancer) may be given during protocol treatment; patients are allowed to have received neoadjuvant and/or adjuvant chemotherapy that was completed at least 6 months prior to registration to the protocol
* Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/ social situations that would limit compliance with study requirements
* Patients with known allergy to mushrooms

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01-29 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Feasibility and toxicity of this regimen at six different dose levels | 1 year after treatment on study

SECONDARY OUTCOMES:
Effect on testosterone, dihydrotestosterone, dehydroepiandrosterone, estrogens, aromatase, parameters of the immune function, and circulating tumor cells | 1 year after treatment on study
Effect on PSA kinetics | 1 year after treatment on study

CONTACTS AND LOCATIONS:
Overall Officials: Cy Stein, MD, PhD, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, South Pasadena, California

REFERENCES:
- [Derived] Twardowski P, Kanaya N, Frankel P, Synold T, Ruel C, Pal SK, Junqueira M, Prajapati M, Moore T, Tryon P, Chen S. A phase I trial of mushroom powder in patients with biochemically recurrent prostate cancer: Roles of cytokines and myeloid-derived suppressor cells for Agaricus bisporus-induced prostate-specific antigen responses. Cancer. 2015 Sep 1;121(17):2942-50. doi: 10.1002/cncr.29421. Epub 2015 May 18. PMID 25989179